CLINICAL TRIAL: NCT03586882
Title: Effect of Spinal Cord Stimulation on Gait and Balance in Chronic Low Back Pain Patients With or Without Leg Pain
Brief Title: Effect of Spinal Cord Stimulation on Gait and Balance in Chronic Low Back Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Texas Back Institute (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TBIRF-Medt
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-06

CONDITIONS: Chronic Low Back Pain; Pain in Leg, Unspecified
MeSH Terms: interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Spinal Cord Stimulation Group (Experimental): Gait and balance testing as well as self-reported outcome assessments to be administered before and after surgery
  Interventions: Device: Spinal Cord Stimulation
- Control Group (No Intervention): Gait and balance testing to be administered once in healthy subjects

INTERVENTIONS:
Device: Spinal Cord Stimulation — Stimulation provided by the generator to electrodes on the leads inhibits ascending pain signals, thereby decreasing pain perception.
  Arms: Spinal Cord Stimulation Group

SUMMARY:
Spinal Cord Stimulation (SCS) uses electrical signals to disrupt noxious signals arising from painful areas, thereby reducing pain perception. Successful SCS implants lead to a broad range of positive outcomes: 1) long-term pain can be expected to be reduced by at least by 50%; 2) quality of life as assessed by subjective measurements improves substantially; 3) patients can significantly reduce opioid medication intake.1 However, the impacts of SCS intervention on neuromuscular and biomechanical outcomes including gait and balance have not been fully explored. Fifty subjects with symptomatic leg pain and/or low back pain (LBP) who are deemed appropriate SCS candidates and are scheduled for surgery will undergo gait and balance analyses preoperatively as well as 6 weeks and 3 months post operatively. In addition, 50 control subjects having no pain will undergo 1 session of gait and balance assessment. Objective spine and lower extremity motion and neuromuscular control will be evaluated using dynamic surface EMG and a video motion capture system during functional evaluation. Also, explored will be the relationship of changes in gait and balance to psychosocial factors that have previously been shown to be correlated with SCS outcomes.

DETAILED DESCRIPTION:
Low back pain is reported in 75-80% of the population and can significantly influence patients' quality of life. Fortunately, 80-90% of individuals recover from their back pain, whether they receive treatment or not. However, the small percentage of people who do not recover quickly present a costly problem to society and a great challenge to health care providers. Low back pain is the second leading cause for missed days at work, potentially having disability and major socioeconomic consequences. Chronic LBP can also limit flexibility and/or range of motion, which may contribute to an overall decrease in functional capacity, and may ultimately heighten the risk for additional lower extremity injury. Many chronic LBP patients have conditions not amenable to spine surgery, or they have failed to achieve successful outcome with previous spine surgery. For these patients, SCS can be an effective alternative. For example, in a recent demonstration, randomized 100 failed back surgery syndrome (FBSS) patients to either SCS or conventional medical management. At 6 months post-implant, 64% of patients had achieved the 50% reduction in leg pain criterion (vs. 18% of conventional medical management patients). Similarly, North et al. found 52% of patients had achieved at least the 50% reduction in pain when they investigated 171 patients treated with SCS.

SCS uses electrical signals to decrease nociception of impulses arising from painful areas in the spine and or leg. In order to accomplish this goal, SCS involves implantation of a small electrical pulse generator, along with thin leads strategically placed into the epidural space. Stimulation provided by the generator to electrodes on the leads inhibits ascending pain signals, thereby decreasing pain perception. Occasionally, some patients feel a mild paresthesia as a result of the stimulation.

While the effectiveness of SCS on reduction of subjective pain complaints is now well-established, such improvement may not translate into improved functional ability. Previous research found that, for FBSS patients treated with SCS, patients' scores on Oswestry Disability index did not correlate significantly with improvements in function as measured by an accelerometer contained within the stimulator device. Very few studies have examined the effect of SCS on objectively-measured functional abilities, including gait and balance. Those studies suffer from a small sample size and lack of electromyography (EMG) and full body kinematics analyses. Despite that, those studies did find improvement in the spatiotemporal variables (i.e. gait speed, step length and width) while other variables (ground reaction force and trunk motion) were not significantly different using the SCS.

Therefore, the purpose of this study is to evaluate the effect of SCS, on the biomechanics of the lower extremities and spine, using dynamic EMG, video motion capture, and force plate analysis, during gait and static balance testing, in patients with chronic low back and/or leg pain, before and after intervention. In addition this study will compare these same biomechanical parameters found in the chronic low back pain and /or leg pain patients to an asymptomatic control group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Considered to be a candidate for SCS

   1. Leg pain and/or LBP lasting than 6 months.
   2. Therapy consists of a short trial with a percutaneous implantation of neurostimulator electrode(s) in the epidural space for assessing a candidate's suitability for ongoing treatment with a permanent surgically implanted SCS. Performance and documentation of an effective trial is required for consideration of permanent SCS.
   3. The implantation of the stimulator is used only as a late or last resort for patients with chronic intractable pain.
   4. Other treatment modalities (pharmacologic, surgical, physical/and psychological therapies) have been tried and did not prove satisfactory; were judged unsuitable, or were contraindicated for the patient.
   5. Patient has undergone appropriate psychological screening, including psychometric testing using the Minnesota Multiphasic Personality Inventory-2 Restructured Form (MMPI-2-RF), and diagnosis by a multidisciplinary team before implantation; to include patient education, discussion and disclosure including an extensive discussion of the risk and benefits of therapy.
   6. All the facilities, equipment, and professional support personnel required for the proper diagnosis, treatment, training, and follow-up of the patient are available.
   7. All trials which proceed to permanent implantation should demonstrate adequate documentation to support the decision. A successful trial should be associated with at least 50% reduction of target pain, a reduction of analgesic medications and show some element of functional improvement (i.e. sitting, standing and walking tolerances).
3. Able to ambulate without assistance and stand without assistance with eyes open for a minimum of 10 seconds
4. Able and willing to attend and perform the activities described in the informed consent within the boundaries of the timelines set forth for pre-, and post-operative follow-up

Exclusion Criteria:

1. Major lower extremity surgery or previous injury that may affect gait (a successful total joint replacement is not an exclusion)
2. BMI higher than 35
3. Neurological disorder, diabetic neuropathy or other disease that impairs the patient's ability to ambulate or stand without assistance
4. Major trauma to the pelvis
5. Pregnant or wishing to become pregnant during the study
6. Previous spinal surgery that would preclude the safe percutaneous or permanent implantation of the SCS leads
7. Previous history of spinal infection either iatrogenic or denovo
8. Previous SCS attempts either successful or not

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Kinematic Variables Change assessed with human motion capture system | Baseline; 6 and 12 weeks after surgery
  3-Dimensional Range of Motion (ROM) during the stance and swing phase of the spine, pelvis, hip, knee, ankle, shoulder, and elbow joint angles along with center of mass and head sway and displacement

SECONDARY OUTCOMES:
Patient Self-Reported Outcome Assessments Change - Visual analog scale (VAS) | Baseline; 6 and 12 weeks after surgery
  VAS for lower back pain, neck and arm pain, and leg pain. Scale range from 0 (no pain) - 10 (most pain)
Patient Self-Reported Outcome Assessments Change - Oswestry Disability Index (ODI, version 2.1.a). | Baseline; 6 and 12 weeks after surgery
  Scale range from 0 (no pain) - 10 (most pain)
Patient Self-Reported Outcome Assessments Change - Tampa Scale for Kinesiophobia (TSK). | Baseline; 6 and 12 weeks after surgery
  TSK is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement.
Patient Self-Reported Outcome Assessments Change - Minnesota Multiphasic Personality Inventory - 2 - Restructured Form (MMPI-2-RF). | Baseline; 6 and 12 weeks after surgery
  The MMPI-2-RF is a 338-item, self-report inventory that assesses personality and psychopathology across 42 substantive scales.

OTHER OUTCOMES:
Kinetic Variables Change assessed with human motion capture system | Baseline; 6 and 12 weeks after surgery
  Vertical Ground Reaction Forces (GRF)
Spatio-Temporal Variables Change assessed with human motion capture system | Baseline; 6 and 12 weeks after surgery
  Walking speed
Neuromuscular Variables Change assessed with an Electromyography | Baseline; 6 and 12 weeks after surgery
  Bilateral peak magnitude during the stance phase

CONTACTS AND LOCATIONS:
Overall Officials: Ram Haddas, PhD, Principal Investigator — Texas Back Institute
Locations (1):
- Texas Back Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gee L, Smith HC, Ghulam-Jelani Z, Khan H, Prusik J, Feustel PJ, McCallum SE, Pilitsis JG. Spinal Cord Stimulation for the Treatment of Chronic Pain Reduces Opioid Use and Results in Superior Clinical Outcomes When Used Without Opioids. Neurosurgery. 2019 Jan 1;84(1):217-226. doi: 10.1093/neuros/nyy065. PMID 29538696
- [Background] Waddell G. 1987 Volvo award in clinical sciences. A new clinical model for the treatment of low-back pain. Spine (Phila Pa 1976). 1987 Sep;12(7):632-44. doi: 10.1097/00007632-198709000-00002. PMID 2961080
- [Background] Block AR, Gatchel RJ, Deardorff WW, et al. The Psychology of Spine Surgeryed. Washington, D.C.: American Psychological Association, 2003.
- [Background] Frey ME, Manchikanti L, Benyamin RM, Schultz DM, Smith HS, Cohen SP. Spinal cord stimulation for patients with failed back surgery syndrome: a systematic review. Pain Physician. 2009 Mar-Apr;12(2):379-97. PMID 19305486
- [Background] Mekhail NA, Mathews M, Nageeb F, Guirguis M, Mekhail MN, Cheng J. Retrospective review of 707 cases of spinal cord stimulation: indications and complications. Pain Pract. 2011 Mar-Apr;11(2):148-53. doi: 10.1111/j.1533-2500.2010.00407.x. Epub 2010 Sep 8. PMID 21371254
- [Background] Eldabe S, Kumar K, Buchser E, Taylor RS. An analysis of the components of pain, function, and health-related quality of life in patients with failed back surgery syndrome treated with spinal cord stimulation or conventional medical management. Neuromodulation. 2010 Jul;13(3):201-9. doi: 10.1111/j.1525-1403.2009.00271.x. Epub 2010 Feb 22. PMID 21992833
- [Background] Agari T, Date I. Spinal cord stimulation for the treatment of abnormal posture and gait disorder in patients with Parkinson's disease. Neurol Med Chir (Tokyo). 2012;52(7):470-4. doi: 10.2176/nmc.52.470. PMID 22850494
- [Background] Turner JA, Hollingworth W, Comstock BA, Deyo RA. Spinal cord stimulation for failed back surgery syndrome: outcomes in a workers' compensation setting. Pain. 2010 Jan;148(1):14-25. doi: 10.1016/j.pain.2009.08.014. Epub 2009 Oct 28. PMID 19875232
- [Background] de Andrade DC, Bendib B, Hattou M, Keravel Y, Nguyen JP, Lefaucheur JP. Neurophysiological assessment of spinal cord stimulation in failed back surgery syndrome. Pain. 2010 Sep;150(3):485-491. doi: 10.1016/j.pain.2010.06.001. Epub 2010 Jun 29. PMID 20591571
- [Background] North RB, Kidd DH, Zahurak M, James CS, Long DM. Spinal cord stimulation for chronic, intractable pain: experience over two decades. Neurosurgery. 1993 Mar;32(3):384-94; discussion 394-5. doi: 10.1227/00006123-199303000-00008. PMID 8455763
- [Background] Geurts JW, Joosten EA, van Kleef M. Current status and future perspectives of spinal cord stimulation in treatment of chronic pain. Pain. 2017 May;158(5):771-774. doi: 10.1097/j.pain.0000000000000847. No abstract available. PMID 28106667
- [Background] Goudman L, Smet I, Marien P, De Jaeger M, De Groote S, Huysmans E, Putman K, Van Buyten JP, Buyl R, Moens M. Is the Self-Reporting of Failed Back Surgery Syndrome Patients Treated With Spinal Cord Stimulation in Line With Objective Measurements? Neuromodulation. 2018 Jan;21(1):93-100. doi: 10.1111/ner.12719. Epub 2017 Nov 3. PMID 29105225
- [Background] Rijken NH, Vonhogen LH, Duysens J, Keijsers NL. The effect of spinal cord stimulation (SCS) on static balance and gait. Neuromodulation. 2013 May-Jun;16(3):244-50; discussion 249-50. doi: 10.1111/j.1525-1403.2012.00512.x. Epub 2012 Sep 25. PMID 23009103
- [Background] Brugliera L, De Luca A, Corna S, Bertolotto M, Checchia GA, Cioni M, Capodaglio P, Lentino C. Spinal Cord Stimulation in Failed Back Surgery Syndrome: Effects on Posture and Gait-A Preliminary 3D Biomechanical Study. Pain Res Manag. 2017;2017:3059891. doi: 10.1155/2017/3059891. Epub 2017 Sep 25. PMID 29147083
- [Background] Al-Kaisy A, Palmisani S, Smith TE, Pang D, Lam K, Burgoyne W, Houghton R, Hudson E, Lucas J. 10 kHz High-Frequency Spinal Cord Stimulation for Chronic Axial Low Back Pain in Patients With No History of Spinal Surgery: A Preliminary, Prospective, Open Label and Proof-of-Concept Study. Neuromodulation. 2017 Jan;20(1):63-70. doi: 10.1111/ner.12563. Epub 2016 Dec 26. PMID 28025843
- [Background] Sumner LA, Lofland K. Spinal cord stimulation: Subjective pain intensity and presurgical correlates in chronic pain patients. Chronic Illn. 2014 Sep;10(3):157-66. doi: 10.1177/1742395313504233. Epub 2013 Sep 18. PMID 24048947
- [Background] Wolter T, Kieselbach K. Cervical spinal cord stimulation: an analysis of 23 patients with long-term follow-up. Pain Physician. 2012 May-Jun;15(3):203-12. PMID 22622904
- [Background] Vaughan CL, Davis BL, O'Conner JC. Dynamics of Human Gait. 2nd ed. Cape Town, South Africa: Kiboho Publishers, 1999.
- [Background] Arumugam A, Milosavljevic S, Woodley S, Sole G. Effects of external pelvic compression on form closure, force closure, and neuromotor control of the lumbopelvic spine--a systematic review. Man Ther. 2012 Aug;17(4):275-84. doi: 10.1016/j.math.2012.01.010. Epub 2012 Mar 2. PMID 22386280
- [Background] Lethem J, Slade PD, Troup JD, Bentley G. Outline of a Fear-Avoidance Model of exaggerated pain perception--I. Behav Res Ther. 1983;21(4):401-8. doi: 10.1016/0005-7967(83)90009-8. No abstract available. PMID 6626110
- [Background] Miller RP, Kori S, Todd D. The Tampa Scale: a measure of kinesiophobia. Clin J Pain 1991;7:51-2.
- [Background] Lundberg MKE, Styf J, Carlsson SG. A psychometric evaluation of the Tampa Scale for Kinesiophobia - from a physiotherapeutic perspective. Physiotherapy Theory and Practice 2004;20:121-33.
- [Background] Lundberg M, Styf J, Jansson B. On what patients does the Tampa Scale for Kinesiophobia fit? Physiother Theory Pract. 2009 Oct;25(7):495-506. doi: 10.3109/09593980802662160. PMID 19925172
- [Background] Bunketorp L, Carlsson J, Kowalski J, Stener-Victorin E. Evaluating the reliability of multi-item scales: a non-parametric approach to the ordered categorical structure of data collected with the Swedish version of the Tampa Scale for Kinesiophobia and the Self-Efficacy Scale. J Rehabil Med. 2005 Sep;37(5):330-4. doi: 10.1080/16501970510036411. PMID 16208869
- [Background] Wertli MM, Rasmussen-Barr E, Weiser S, Bachmann LM, Brunner F. The role of fear avoidance beliefs as a prognostic factor for outcome in patients with nonspecific low back pain: a systematic review. Spine J. 2014 May 1;14(5):816-36.e4. doi: 10.1016/j.spinee.2013.09.036. Epub 2013 Oct 18. PMID 24412032
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Rainville J, Smeets RJ, Bendix T, Tveito TH, Poiraudeau S, Indahl AJ. Fear-avoidance beliefs and pain avoidance in low back pain--translating research into clinical practice. Spine J. 2011 Sep;11(9):895-903. doi: 10.1016/j.spinee.2011.08.006. Epub 2011 Sep 9. PMID 21907633
- [Background] Ben-Porath YS, Tellegen A. MMPI-2-RF Manual for Administration, Scoring, and Interpretationed. Minneapolis, MN: University of Minnesota Press, 2008.
- [Background] Block AR, Marek RJ, Ben-Porath YS, Kukal D. Associations Between Pre-Implant Psychosocial Factors and Spinal Cord Stimulation Outcome: Evaluation Using the MMPI-2-RF. Assessment. 2017 Jan;24(1):60-70. doi: 10.1177/1073191115601518. Epub 2015 Aug 28. PMID 26318387
- [Background] Block AR, Ben-Porath YS, Marek RJ. Psychological risk factors for poor outcome of spine surgery and spinal cord stimulator implant: a review of the literature and their assessment with the MMPI-2-RF. Clin Neuropsychol. 2013;27(1):81-107. doi: 10.1080/13854046.2012.721007. Epub 2012 Sep 21. PMID 22998432